CLINICAL TRIAL: NCT05713851
Title: Potential Use of Dapaglifozin to Avoid Acute Kindey Injury (AKI) to Chronic Kidney Disease (CKD) Transition: DAKI-CKD Study
Brief Title: Dapaglifozin to Avoid Acute Kindey Injury (AKI) to Chronic Kidney Disease (CKD) Transition: DAKI-CKD Study
Acronym: DAKI-CKD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Olynka Vega Vega (Unknown); Noemi del Toro Cisneros (Unknown); Miguel Ángel Martínez Rojas (Unknown)
Responsible Party: Principal Investigator, Norma Bobadilla, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4301
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: AKI - Acute Kidney Injury; Biomarkers; Transition to CKD; CKD
Keywords: AKI; Biomarkers; no recovery
MeSH Terms: conditions — Acute Kidney Injury | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Group 1: Dapagliflozin 10 mg, will be administered orally or by nasogastric tube every 24 h for 21 days.
  Group 2: Standard of care strategy, patients will receive the usual treatment for their pathology according to the judgment of their treating physician and the Institutional practices, without receiving any of the interventional drugs, but blood and urinary samples will be taken to determine the biomarkers at the times established in the schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapaglifozin group (Experimental): Dapagliflozin 10 mg, will be administered orally or by nasogastric tube every 24 h for 21 days.
  Interventions: Drug: Dapagliflozin
- Standard of care (Placebo Comparator): Without receiving any of the interventional drugs.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — dapagliflozin is given for 21 days vs standard of care

SUMMARY:
Justification: Studies in recent years have shown that suffering an episode of acute kidney injury (AKI) is an independent risk factor for developing chronic kidney disease (CKD), which is associated with cardiovascular complications, increases medical care costs, and decreases survival. These AKI to ERC transition cases add to the growing number of CKD cases already being seen globally. It is for them that in recent years therapeutic strategies have been sought to reduce or stop this process of transition from AKI to CKD.

Objective: To evaluate the efficacy and safety of the use of dapagliflozin plus standard medical treatment (TMS), compared with only TMS for 21 days, in hospitalized patients with a diagnosis of severe AKI (KDIGO 3) in reducing the incidence of CKD to 18 months of follow-up.

Design: Randomized, single center, open study. 100 hospitalized patients with a diagnosis of AKI KDIGO 3, without previous CKD, will be randomized to receive 10 mg of dapagliflozin every 24 h for 21 days + TMS or only TMS. During their follow-up, baseline blood and urine samples will be taken and at 3, 6, 12 and 18 months. At 18 months, the development of CKD will be assessed using the KDIGO clinical criteria and with the determination of urinary biomarkers (Serpina A3, HSP72, KIM 1 and NGAL).

DETAILED DESCRIPTION:
It is planned to randomize 100 patients, 50 for each arm of the study. The randomization will be 1: 1 based on an open access computer program.

Group 1: Dapagliflozin 10 mg, will be administered orally or by nasogastric tube every 24 h for 21 days.

Group 2: Standard of care strategy, patients will receive the usual treatment for their pathology according to the judgment of their treating physician and the Institutional practices, without receiving any of the interventional drugs.

Eligibility: Adults (aged >18 years) with AKI 3 diagnosis for less than 24 h (KDIGO classification, creatinine level or urine output criteria), hospitalized in general admission floor and/or intensive care unit. AKI diagnosis must be compatible with the diagnosis of acute tubular necrosis in a context of ischemic or toxic aggression.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged >18 years) with AKI 3 diagnosis for less than 24 h (KDIGO classification, creatinine level or urine output criteria), hospitalized in general admission floor and/or intensive care unit. AKI diagnosis must be compatible with the diagnosis of acute tubular necrosis in a context of ischemic or toxic aggression.

Exclusion Criteria:

* CKD Stage 3b (KDIGO) or more, renal transplant, urinary tract obstruction, thrombotic microangiopathy, acute glomerulopathy, cardiac arrest without awakening, oncological diagnosis with a life expectancy of less than 5 years, use of norephinephrine >0.30 mcg/kg/min for 6 h or more, use of two vasopressors, PaO2/FiO2 ratio <150, Type 1 DM, fasting for more than 48 h, previous inclusion in other study, pregnant or breastfeeding woman.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the mean change in urinary Serpin A3 (uSerpinA3) levels 18 months after randomization of the patients. | 18 months

SECONDARY OUTCOMES:
GFR at 18 months of randomization calcutated with CKD-EPI creatinine-Cystatin C Equation. | 18 months
Urine HSP-72 levels 18 months after randomization of the patients | 18 months
Urine NGAL levels 18 months after randomization of the patients | 18 months
Urine KIM-1 levels 18 months after randomization of the patients | 18 months
Serum Cystatin C levels 18 months after randomization of the patients | 18 months
Serum creatinine levels 18 months after randomization of the patients | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
117 / 5,000 Resultados de traducción Traducción star_border Once the patients have been recruited and the analysis has been carried out, the complete data will be made available in a supplement